CLINICAL TRIAL: NCT02027987
Title: Clinical Study on the Neuroprotection and Epilepsy Prevention of Valproate Acid Administered After Severe Traumatic Brain Injury
Brief Title: Traumatic Neuroprotection and Epilepsy Prevention of Valproate Acid
Acronym: VPA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20130814-7
Record Dates: First submitted 2013-10-28; First posted 2014-01-06 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2013-11

CONDITIONS: Traumatic Brain Injury
Keywords: valproate acid; traumatic brain injury; brain protection; epilepsy
MeSH Terms: conditions — Brain Injuries, Traumatic; Epilepsy | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- valproate acid (Experimental): The patients began receiving treatment at a dose of 400 mg VPA twice daily on the day after randomization by intravenous drip, with this dose continued for 14 days.The dose was increased to 500 mg twice daily at week 3 and to 400 mg three times daily at week 4 if the DRS score had not improved by at least 2 points from baseline. After the week 4 assessment, the study drug was tapered over a period of 2 to 3 days, with assessment of the patients continued through week 6. Additional procedural details are provided in the study protocol.
  Interventions: Drug: valproate acid
- placebo (Placebo Comparator)

INTERVENTIONS:
Drug: valproate acid — valproate acid is a common drug which is applied for epilepsy prevention and treatment.
  Other Names: Sodium valproate
  Arms: valproate acid

SUMMARY:
1. Background:

   Preliminary studies have suggested that valproate acid (VPA) may promote neuron survival, inhibit apoptosis, decrease the neuron function deficit in cerebral ischemia, and promote the brain functional recovery after traumatic brain injury (TBI). Besides, in the guide of prevention and treatment of epilepsy in 2007, VPA was one of the antiepileptic drugs which were suggested to prevent early epilepsy after TBI (less than 7 days).
2. Objectives:

   Our main objective was to evaluate whether VPA could protect brain and improve recovery of brain function after severe TBI. The secondary objective was to explore whether VPA could prevent late epilepsy after severe TBI (more than 7 days).
3. Methods:

We would enroll 160 patients who were in a vegetative or minimally conscious state 4 to 16 weeks after TBI and who were receiving inpatient rehabilitation. Patients were randomly assigned to receive VPA or placebo for 4 weeks and were followed for 2 weeks after the treatment was discontinued. The rate of functional recovery on the Disability Rating Scale (DRS; range, 0 to 29, with higher scores indicating greater disability) was compared over the 4 weeks of treatment (primary outcome) and during the 2-week washout period with the use of mixed-effects regression models.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were 16 to 65 years of age with all genders.
* The patients had sustained a nonpenetrating traumatic brain injury 4 to 16 weeks before enrollment, with the confirmation of CT or MRI.
* Additional eligibility criteria were a vegetative state or a minimally conscious state, as indicated by a Disability Rating Scale (DRS) score greater than 11.
* There was an inability both to follow commands consistently and to engage in functional communication, as assessed by the score on the Coma Recovery Scale-Revised (CRS-R)
* All the patients had provided written informed consent.
* The patients were receiving usual inpatient rehabilitation and treatment at each site.

Exclusion Criteria:

* unstable health state,including:Be allergic to VPA, or with serious allergic diseases or allergic constitutions;With serious cardiovascular diseases, hepatic, renal, or psychiatric diseases;With serious respiratory, endocrine, or blood system diseases;With serious infections or malignant tumors; With weakened immunologic status;Addison's diseases;With alcohol or drug abuse.
* Any disability related to the central nervous system that predated the traumatic brain injury.
* Pregnancy or breastfeeding females.
* More than one seizure in the previous month.
* Prior treatment with VPA
* In the case of patients who were undergoing evaluation for ventricular shunt placement or receiving a psychoactive medication, enrollment was deferred until shunt placement had been completed or psychoactive medications discontinued.
* The patients had enrolled the other studies in the past three months or are engaging the other studies.
* The patients were assessed as unqualified for the study according to the comprehensive evaluation opinion brought forward by the research team.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
DRS scores | On the 0,7th,14th,21st,28th,35th,42nd days since admitted into the study
  The DRS score includes measures of eye opening, verbalization, and motor response (derived from the Glasgow Coma Scale); cognitive understanding of feeding, dressing, and grooming; degree of assistance and supervision required; and employability. Scores range from 0 to 29, with higher values indicating greater disability.

SECONDARY OUTCOMES:
the time of break out and state of epilepsy | from 0 to 42 days when the epilepsy break out
  When the patient were admitted into the study, the breakout and the severity of epilepsy would be monitored and treated until the end of the trial.
brain MRI scan | 6 weeks after treatment
  Brain MRI scan is applied to monitor the degree and progress of the brain damage.
the blood concentration of VPA | On the 0,7th,14th,21st,28th,35th,42nd days since admitted into the study
  the blood was collected to detect the concentration about 2 hours after the medication of VPA

OTHER OUTCOMES:
CRS-R score | On the 0,7th,14th,21st,28th,35th,42nd days since admitted into the study
  The CRS-R score is a standardized neurobehavioral assessment tool comprising six hierarchically organized subscales (i.e., auditory, visual, motor, oromotor-verbal, communication, and arousal); scores range from 0 to 23, with higher scores indicating a higher level of neurobehavioral function.
function of kidney | On the 0,7th,14th,21st,28th,35th,42nd days since admitted into the study
  There are three main indicators: blood creatinine, urea nitrogen, and uric acid. These indicator are used as a monitor of the kidney safety.
function of liver | On the 0,7th,14th,21st,28th,35th,42nd days since admitted into the study
  There are several main indicators including ALT, AST, Tbil, D-bil, I-bil, ALB,GLB, and ALP, and so on. These indicators could monitor the change of liver function in case of liver damage.
Physiological and pathological reflex check | On the 0,7th,14th,21st,28th,35th,42nd days since admitted into the study
muscular strength and tension test | On the 0,7th,14th,21st,28th,35th,42nd days since admitted into the study
  There are 6 grades in muscular strength test. And muscular tension test was referred to Modified Ashworth scale.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Zhou, M.D., Ph.D., Study Director — Institute of Neurosurgery, Xijing Hospital, Fourth Military Medical University
Locations (1):
- Institute of Neurosurgery, Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China